CLINICAL TRIAL: NCT06923423
Title: Effectiveness, Implementation, and Cost of Cognitive Processing Therapy in Prisons
Acronym: STRIDES2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 297770; R01DA059549 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-04-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PTSD - Post Traumatic Stress Disorder; PTSD and Alcohol Use Disorder; PTSD and Trauma-related Symptoms; Substance Use Disorder (SUD); Depression; Mental Health; Trauma; Trauma Exposure; Traumatic Stress Disorder; Traumatic Stress; Post Traumatic Stress Symptoms
Keywords: Post traumatic Stress Disorder; Post traumatic Stress Symptoms; Substance Use; Substance Use Disorder; Cognitive Processing Therapy; Cognitive Processing Therapy for Criminal Justice Setting; Trauma focused self help; Facilitation; Implementation Facilitation; Implementation; Cost Estimation and Offsets; Drug Use Disorder; Alcohol Use Disorder; Trauma; Depression; Adult; Incarcerated; Prison; Imprisonment; Intervention; Treatment Comparison; Acceptability; Feasibility; Budget Impact; Cost Estimate; Implementation Evaluation; Recidivism; Self Help; Workbook; Criminal Justice; Effectiveness; Evidence Based Intervention; CPT; CPT-CJ
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Alcoholism; Substance-Related Disorders; Depression; Psychological Well-Being; Wounds and Injuries; Stress Disorders, Traumatic; Recidivism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Cognitive Processing Therapy (CPT) (Active Comparator): Participants in CPT group therapy will learn about trauma and how to change upsetting thoughts related to it. Participants will attend up to a total of 12 sessions held 1-2x/week for 90 minutes. No more than 10 participants will be in a group. In this study, CPT provided is a version that was adapted for prisons (CPT-CJ).
  Interventions: Behavioral: Group Cognitive Processing Therapy (CPT)
- Individual trauma focused self-help via workbook (Active Comparator): Participants in the trauma-focused self-help therapy will independently read and do practice assignments in a workbook to learn skills to recover from trauma.
  Interventions: Behavioral: Control Group Individual trauma focused self-help via workbook

INTERVENTIONS:
Behavioral: Group Cognitive Processing Therapy (CPT) — Participants in CPT group therapy will learn about trauma and how to change upsetting thoughts related to it. Participants will attend up to a total of 12 sessions held 1-2x/week for 90 minutes. No more than 10 participants will be in a group. In this study, CPT provided is a version that was adapted for prisons.
  Other Names: CPT-CJ
  Arms: Group Cognitive Processing Therapy (CPT)
Behavioral: Control Group Individual trauma focused self-help via workbook — The self-help therapy is a therapy that people do on their own using a workbook. By reading and doing practice assignments in the workbook, people can learn skills to recover from trauma.
  Arms: Individual trauma focused self-help via workbook

SUMMARY:
Addiction and trauma exposure are common among the 5.5 million people (1 in 47 adults) in the U.S. who are in prison or under supervision. About 85% of people in prison have a substance use disorder or are there for a drug-related crime, and many have experienced serious trauma before being incarcerated. Posttraumatic stress symptoms (PTSS) are often a result of trauma and are linked to more severe drug use, higher rates of relapse, and increased crime. PTSS and substance use disorder (SUD) each raise the chances of new arrests for people who are justice-involved, showing that addressing trauma and addiction could help reduce repeat offenses and the costs of incarceration. However, treatments for PTSS are rarely available in prisons, and there is little research on whether providing therapy for PTSS in prison can lower drug use, PTSS, or crime after release.

The goal of this clinical trial is to see if trauma-focused group therapy (CPT) provided while in prison, can help people after release from prison. The therapy has been adapted for use in prisons (CPT-CJ) and will be compared to trauma focused therapy delivered via a self-help workbook

This study will:

* test whether a trauma-focused group therapy (CPT-CJ) can reduce post-incarceration drug and alcohol use, mental health issues, and drug-related crime, compared to trauma-focused self-help,
* evaluate a strategy called implementation facilitation, which helps support the use of this therapy in prisons, and
* measure the cost of the therapies and support strategies to help plan for future expansion.

Incarcerated participants (N = 640; 50% female) will be enrolled from ~10 prisons in ~5 states, ensuring variability in population and setting characteristics. They will:

* take surveys and answer questions up to 5 times (before starting treatment, right after getting treatment, right before leaving prison, 3 months after leaving prison and 6 months after leaving prison)
* complete CPT group therapy or self-help therapy
* provide urine samples 3 months and 6 months after leaving prison

Prison stakeholders (e.g., prison staff, prison leadership, governmental officials; N = ~15 per site) who will be purposively sampled based on their role in CPT-CJ implementation will also participate in some surveys.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to understand and speak English
* Able to give informed consent
* All items listed in "Inclusion criteria for all participants"
* Be currently incarcerated in one of the prisons that have partnered as study sites
* Have met criteria for a drug use disorder in the year prior to their current incarceration (≥ 2 symptoms on a DSM-5 drug use disorder checklist)
* Have used drugs in the 30 days prior to their current incarceration
* Have a history of traumatic event exposure
* Endorse clinically significant posttraumatic stress symptoms (score ≥ 4 on the Primary Care PTSD Screen for DSM-5; PC-PTSD-5)
* Expect to be incarcerated for at least long enough to complete CPT-CJ as it is being implemented at the particular site (i.e., anticipated to be ~3 months, but will depend on dates associated with next available intervention group)
* Expect to be released from prison within 12 months following the end of treatment (i.e., within ~15 months of the pre-treatment assessment)
* Willing to consent to randomization to treatment condition

Exclusion criteria for prisoners (additional requirements assessed during pre-treatment assessments or indicated by prison staff; will result in being withdrawn from the study prior to randomization by the PI):

* Unable to provide any locator information for post-release assessments
* Determined to be releasing sooner than would allow the individual to complete CPT-CJ
* Determined to have an unavoidable scheduling conflict or facility restriction (e.g., disciplinary, medical) that would prevent participation in CPT-CJ. Of note, if the scheduling conflict or facility restriction is expected to resolve following the next round of randomization at the study site, the participant may be put on "hold for next round" status rather than withdrawn unless other exclusionary criteria would be met by that time (e.g., release).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Drug Use Frequency (Count) | 3- and 6-month post-release from prison
  Participants complete a Timeline Follow Back Interview assessment of illicit drug use during the previous 30 days at 3- & 6-months post-release from prison. The total number of days of drug use will be summed to represent drug use frequency.
Drug use (Binary) | 3- and 6-month post-release from prison
  Participants complete a Timeline Follow Back Interview assessment of illicit drug use during the previous 30 days at 3- & 6-months post-release from prison. The total number of days of drug use will be dichotomized to indicate presence or absence of drug use since release.
Posttraumatic Stress Symptom Severity (Sum) | Pre-treatment assessments will be ~2 wks before tx starts; post-treatment will be ~2 wks after tx ends; pre-release will be ~3 days before release; post-release follow-ups will be 3- and 6-mo after prison exist
  Participants complete the PTSD Checklist for DSM-5 (PCL-5) at all assessments to examine change the effectiveness of the intervention and control groups on posttraumatic stress symptom severity. Scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
Treatment fidelity (ratio) | Fidelity assessments will be done during the active treatment period which can be as short as 6 weeks to as long as 3 months for participants. The active treatment period is expected to span 1.5 years at each site.
  The ratio of the number of CPT-CJ components delivered to the number of CPT-CJ components planned per completed fidelity monitoring templates.

SECONDARY OUTCOMES:
Drug Use Disorder Symptom Severity (Count) | 3- and 6-months post-release from prison
  Participants will complete a DSM-5 checklist of drug use disorder diagnostic criteria. The checklist can result in a maximum score of 11, with scores of 2 or greater indicating the presence of symptoms likely to meet diagnostic criteria. Scores will represent the total number of symptoms currently endorsed.
Drug Use Disorder (Binary) | 3- and 6-months post-release from prison
  Participants will complete a DSM-5 checklist of drug use disorder diagnostic criteria. The checklist can result in a maximum score of 11, with scores of 2 or greater indicating the presence of symptoms likely to meet diagnostic criteria. Scores will represent the total number of symptoms currently endorsed. Sum score will be used to determine substance use disorder presence (i.e., scores ≥ 2) or absence (scores of 0-1).
Depressive Symptom Severity (Sum) | Pre-treatment assessments will be done ~2 wks before tx starts; post-treatment will be ~2 wks after tx ends; pre-release will be ~3 days before release; post-release follow-ups will be ~3- and ~6-mo after prison exit
  Participants will complete the Patient Health Questionnaire - 8-item (PHQ-8) at all assessments to examine change the effectiveness of the intervention and control groups on depressive symptom severity. Scores range from 0-24 with higher scores indicating more severe depressive symptoms.
Alcohol Use Frequency (Count) | 3- and 6-months post-release from prison
  Participants will complete a Timeline Follow Back Interview assessment of alcohol use during the previous 30 days at both 3- and 6-months post-release from prison. The total number of days of alcohol use will be summed to represent drug use frequency.
Alcohol Use (Binary) | 3- and 6-months post-release from prison
  Participants will complete a Timeline Follow Back Interview assessment of alcohol use during the previous 30 days at both 3- and 6-months post-release from prison. The total number of days of alcohol use will be dichotomized to indicate presence or absence of alcohol use since release.
Alcohol Use Disorder Symptom Severity (Count) | 3- and 6-months post-release from prison
  Participants will complete a DSM-5 checklist of alcohol use disorder diagnostic criteria. The checklist can result in a maximum score of 11, with scores of 2 or greater indicating the presence of symptoms likely to meet diagnostic criteria. Scores will represent the total number of symptoms currently endorsed.
Alcohol Use Disorder (Binary) | 3- and 6-months post-release from prison
  Participants will complete a DSM-5 checklist of alcohol use disorder diagnostic criteria. The checklist can result in a maximum score of 11, with scores of 2 or greater indicating the presence of symptoms likely to meet diagnostic criteria. Scores will represent the total number of symptoms currently endorsed. Sum score will be used to determine substance use disorder presence (i.e., scores ≥ 2) or absence (scores of 0-1).
Drug-Related Crime Frequency (Count) | 6-months post-release from prison
  Sum of new arrests and new convictions for drug charges based on the Criminal and Legal Activities Form and, if sufficient data is available, administrative records.
Drug Related Crime (Binary) | 6-months post-release from prison
  Presence or absence of any new arrests or new convictions for drug charges based on the Criminal and Legal Activities Form and, if sufficient data is available, administrative records.
Substance-Related Disciplinary Violations (Count) | Interval between treatment completion and release from incarceration, which could be as short as 1 day and as long as ~2 years
  Sum of substance-related disciplinary violations received while incarcerated per administrative records
Substance-Related Disciplinary Violations (Binary) | Interval between treatment completion and release from incarceration, which could be as short as 1 day and as long as ~2 years
  Presence or absence of any substance-related disciplinary violations received while incarcerated per administrative records.
Positive Urine Drug Screens (Binary) | 3- and 6-months post-release from prison
  Presence or absence of any positive urine drug screens following release from prison per department of corrections administrative records.
Treatment Acceptability (mean) | Post-treatment assessments will be completed 2 weeks after treatment ends (for residents). Immediately and 12-months post-implementation (for prison stakeholders)
  Prison residents and stakeholders will complete the Acceptability of Intervention Measure (AIM) to index treatment acceptability. Mean scores on the AIM range from 1-5, with higher scores indicating greater intervention acceptability.
Treatment Acceptability (sum) | Administered at post-treatment assessment, which will be completed ~2 weeks after treatment ends
  Prison residents will complete the Client Satisfaction Questionnaire (CSQ-8) as an additional index of treatment acceptability. Sum scores on the CSQ-8 range from 8-32, with higher scores indicating greater intervention acceptability.
Treatment appropriateness (mean) | Post-treatment assessments will be completed ~2 weeks after treatment ends (for residents). Immediately and 12-months post-implementation (for prison stakeholders)
  The Intervention Appropriateness Measure (IAM) will be completed by both prison residents and prison stakeholders. Mean scores on the IAM range from 1-5, with higher scores indicating greater intervention appropriateness.
Treatment feasibility (mean) | Immediately and 12-months post-implementation
  The Feasibility of Intervention Measure (FIM) will be completed by prison stakeholders to index treatment feasibility. Mean scores on the FIM range from 1-5, with higher scores indicating greater intervention feasibility.
Treatment adoption (ratio) | Treatment adoption assessment will be done during the active treatment period, which can be as short as 6 weeks to as long as 3 months for participants. The active treatment period is expected to span 1.5 years at each site
  Ratio of patients who completed CPT-CJ to the number who were randomized
Treatment sustainability (ratio) | 1-year post-implementation
  The number of sites of total that are maintaining or increasing in CPT-CJ provision with high fidelity after implementation facilitation support is withdrawn.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Zielinski, PhD, Principal Investigator — University of Arkansas
Locations (6):
- United States (6):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Northeast Arkansas Community Corrections Center (NEACC), Osceola, Arkansas
  - Southwest Arkansas Community Correction Center, Texarkana, Arkansas
  - East Central Arkansas Community Correction Center, West Memphis, Arkansas
  - North Dakota State Penitentiary (NDSP), Bismarck, North Dakota
  - Heart River Correctional Center (HRCC), Bismarck, North Dakota

IPD SHARING:
Plan to Share IPD: Undecided